CLINICAL TRIAL: NCT02290691
Title: Inactivated Influenza Via Jet Injection
Acronym: IIJI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PharmaJet, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PJ-501-14
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Results first posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Influenza, Human
Keywords: Needle Free, Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Needle- Free (Experimental): Subjects will receive a single 0.5mL injection of inactivated influenza vaccine in the deltoid region on Day 0.
  Interventions: Biological: Influenza Vaccine
- Needle and Syringe (Active Comparator): Subjects will receive a single 0.5mL injection of inactivated Influenza Vaccine in the deltoid region on Day 0.
  Interventions: Biological: Influenza Vaccine

INTERVENTIONS:
Biological: Influenza Vaccine — Influenza Vaccine

SUMMARY:
The purpose of this study is to determine if the administration of flu vaccine using Needle-Free is equivalent to Needle and Syringe administration as measured by laboratory tests of immune response.

DETAILED DESCRIPTION:
Primary:

To evaluate the non-inferiority of flu vaccine administered by needle-free intramuscular (IM) injection versus needle and syringe IM injection as determined with serum hemagglutination inhibition (HAI) reciprocal titers in healthy adults between 18-64 years.

Secondary:

To compare tolerability and safety of the vaccine in the same population based on specifically solicited local and systemic reactions occurring through 7 days post-immunization and adverse events spontaneously reported through approximately 28 days post immunization.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 and ≤ 64 years of age at time of enrollment
* Willing and able to give informed consent after reading the consent form and given adequate opportunity to discuss the study with the investigator or qualified designee
* Willing and able to adhere to all protocol required study procedures and to attend scheduled visits
* Able to receive the trivalent influenza vaccine (TIV) or quadrivalent influenza vaccine (QIV) based on PI judgment
* Stable health status with no exclusionary medical or neuropsychiatric conditions as determined during the screening evaluation and based on the clinical judgment of the investigator or qualified designee
* Access to a consistent means of telephone contact

Exclusion Criteria:

* Presence of any febrile illness (oral temperature >38 °C) on the day of immunization. Such subjects will be reevaluated for enrollment after resolution of illness
* Presence of significant acute or chronic uncontrolled medical or neuropsychiatric illness and /or presence of any significant condition that may prohibit inclusion as determined by the investigator or his qualified designee. Uncontrolled is defined as: requiring institution of a new treatment within 1 month prior to study enrollment or change in medication dosage in the month prior to study enrollment
* Any known immunosuppressive condition including: history of human immunodeficiency virus (HIV) infection, cancer or cancer treatment within 3 years of study enrollment, systemic glucocorticoids (in a dose ≥10 mg prednisone daily or equivalent for more than 7 consecutive days or for 10 or more days in total) within 1 month of study enrollment, or any other cytotoxic or immunosuppressive drug within 3 months of study enrollment. Any significant disorder of coagulation that would increase the risk of intramuscular injections or treatment with Coumadin derivatives or heparin
* Known or suspected to be allergic to eggs, chicken protein, neomycin, polymyxin or influenza vaccine
* History of severe or previous serious adverse reaction after an influenza vaccination
* Receipt of any immunoglobulin and/or blood products within 3 months of immunization or planned administration of any of these products during the study period
* Prior history of any demyelinating disease including Guillain-Barre syndrome.
* Presence of an active neurological disorder
* History of significant alcohol or drug abuse within one year prior to study enrollment
* Influenza vaccination or laboratory confirmed influenza infection within the previous six months before study vaccination or planned influenza vaccination during the study period
* Planned administration of any non-influenza vaccines 30 days prior to the study or during the study period
* Pregnant or plans to become pregnant during the study period
* Currently enrolled in another vaccine or drug study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 985 (Actual)
Dates: Start 2014-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Gannon, MD, Study Director — PharmaJet, Inc.
Locations (6):
- United States (6):
  - Optimal Research LLC, Huntsville, Alabama
  - Optimal Research, LLC, San Diego, California
  - Optimal Research, LLC, Melbourne, Florida
  - Optimal Research, LLC, Peoria, Illinois
  - Optimal Reserach, LLC, Mishawaka, Indiana
  - Optimal Research, LLC, Rockville, Maryland

REFERENCES:
- [Background] McAllister L, Anderson J, Werth K, Cho I, Copeland K, Le Cam Bouveret N, Plant D, Mendelman PM, Cobb DK. Needle-free jet injection for administration of influenza vaccine: a randomised non-inferiority trial. Lancet. 2014 Aug 23;384(9944):674-81. doi: 10.1016/S0140-6736(14)60524-9. Epub 2014 May 31. PMID 24881803

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 05 November 2014 to 15 January 2015 at six clinical centers in the United States.
Pre-assignment Details: A total of 984 participants who met all inclusion criteria and not of the exclusion criteria were enrolled and vaccinated in the study.
Period: Overall Study
Arm/Group | Needle- Free | Needle and Syringe
Started | 496 | 488
Completed | 488 | 479
Not Completed | 8 | 9
Not completed — Noncompliance | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Needle- Free | Needle and Syringe | Total
Number analyzed (Participants) | 496 | 488 | 984
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 496 | 488 | 984
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 241 | 255 | 496
  Male | 255 | 233 | 488

OUTCOME MEASURES:

1. Primary Outcome: Anti Influenza Hemagglutination Inhibition (HAI) Antibody Geometric Mean Titers (GMT)
Description: The GMT criterion for non-inferiority for the upper limit of the 95% CIs of the GMT ratio (GMT with Needle-Free / GMT with Needle and Syringe) antigen will not exceed 1.5 fold.
Time Frame: 28 Days
Population: Geometric mean titers of antibodies against the hemagglutinin (HA) antigens were assessed in the immunogenicity population.
Measure: Geometric Mean (Standard Deviation); unit: Titers
Arm/Group | Needle and Syringe | Needle- Free
Number analyzed (Participants) | 465 | 473
Titers
  A/ H1N1 Day 0 | 3.80 (1.406) | 3.77 (1.441)
  A H1N1 Day 28 | 5.72 (1.109) | 5.70 (1.103)
  A/H3N2 Day 0 | 4.09 (1.549) | 4.09 (1.527)
  A/H3N2 Day 28 | 6.04 (1.104) | 5.99 (1.129)
  B1 Day 0 | 2.83 (1.128) | 2.94 (1.198)
  B1 Day 28 | 4.27 (1.102) | 4.25 (1.150)
  B2 Day 0 | 2.40 (0.904) | 2.52 (0.909)
  B2 Day 28 | 3.83 (0.978) | 3.78 (1.038)

2. Primary Outcome: The Number of Evaluable Participants Achieving Seroconversion or Significant Increase in Antibody Titer.
Description: Seroconversion is defined as a 4-fold rise in HAI titer in post-immunization serum relative to pre-immunization serum, or if pre-immunization serum had an undetectable titer (<1:10), attainment of a post-immunization titer of ≥1:40.
Time Frame: 28 Days
Population: Seroconversion against the hemagglutinin antigens contained in the vaccine were assessed in the Immunogenicity Population.
Measure: Number; unit: participants
Arm/Group | Needle and Syringe | Needle- Free
Number analyzed (Participants) | 465 | 473
participants
  A/H1N1 | 457 | 461
  A/H3N2 | 456 | 468
  B1 | 326 | 365
  B2 | 177 | 167

3. Secondary Outcome: Percentage of Subjects With Immediate Complaints
Description: The following possible immediate complaints will be solicited following the 30 minute safety observation period post-vaccination: local pain, redness, induration/swelling, itching where the injection was given. The data will be reported as "immediate complaints" and presumed to be related to the test article. Any other symptom experienced at 30 minutes will be recorded as an adverse event.
Time Frame: Day 0
Measure: Number; unit: percentage of participants
Arm/Group | Needle and Syringe | Needle- Free
Number analyzed (Participants) | 487 | 496
percentage of participants | 13.6 | 30.2

4. Secondary Outcome: Percentage of Subjects With Solicited Local or Systemic Adverse Events
Description: vaccine reactogenicity will be collected on a patient-completed diary card daily for seven days post-vaccination. The following adverse events will be solicited on the diary card: injection site pain, injection site tenderness, injection site itching, injection site swelling, injection site redness, injection site bruising, fever, fatigue, headache, nausea, chills, muscle ache.
Time Frame: 7 Days
Population: Data included in the analysis were collected on a 7-Day Diary Card from the safety population and grade >1.
Measure: Number; unit: percentage of subjects
Arm/Group | Needle and Syringe | Needle- Free
Number analyzed (Participants) | 488 | 496
percentage of subjects
  Pain | 33.7 | 48.6
  Tenderness | 46.9 | 65.6
  Itching | 6.9 | 24.3
  Redness | 8.2 | 35.5
  Swelling | 6.7 | 29.8
  Bruising | 4.0 | 10.3
  Headache | 16.0 | 14.8
  Fatigue | 15.1 | 11.9
  Muscle Ache | 21.6 | 20.3
  Chills | 6.3 | 4.9
  Nausea | 6.3 | 4.1
  Vomiting | 1.9 | 1.0

5. Secondary Outcome: Percentage of Subjects With Spontaneously Reported Adverse Events
Description: Subjects will be asked to report any other symptoms experienced in addition to the solicited "immediate" and "vaccine reactogenicity" events. Any other events reported will be tabulated as spontaneously reported adverse events.
Time Frame: 28 days
Measure: Number; unit: percentage of subjects
Arm/Group | Needle and Syringe | Needle- Free
Number analyzed (Participants) | 488 | 496
percentage of subjects | 26.5 | 24.4

ADVERSE EVENTS:
Time Frame: Adverse events are reported based on participant recall of events over 28 days
Description: Spontaneously reported adverse events
Arm/Group | Needle- Free | Needle and Syringe
All-Cause Mortality (participants affected / at risk) | 0/496 | 0/488
Serious Adverse Events (participants affected / at risk) | 1/496 | 0/488
Other Adverse Events (participants affected / at risk) | 486/496 | 475/488
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Needle- Free (N=496) | Needle and Syringe (N=488)
influenza and pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Needle- Free (N=496) | Needle and Syringe (N=488)
Pain (General disorders) | 236 (236) | 160 (160)
Tenderness (General disorders) | 319 (319) | 223 (223)
Itching (General disorders) | 118 (118) | 33 (33)
Redness (General disorders) | 173 (173) | 39 (39)
Swelling (General disorders) | 145 (145) | 32 (32)
Bruising (General disorders) | 50 (50) | 19 (19)
Fever (General disorders) | 3 (3) | 9 (9)
Headache (General disorders) | 72 (72) | 76 (76)
Fatigue (General disorders) | 58 (58) | 72 (72)
Muscle Ache (General disorders) | 99 (99) | 103 (103)
Chills (General disorders) | 24 (24) | 30 (30)
Nausea (General disorders) | 20 (20) | 30 (30)
Vomiting (General disorders) | 5 (5) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor may invite Study's Investigators to participate in the preparation of a multicenter article for a professional journal; terms will be at the discretion of the sponsor. Investigators may also wish to publish, present, or use for instruction and research the results of the Study collected at their individual research sites only after publication of pooled, multicenter results and under the following conditions. Materials will be provided to Sponsor for approval prior to submission.